CLINICAL TRIAL: NCT06861439
Title: Effects of Tirzepatide on Fat-Free Mass, Bone and Physical Function in Older Adults - a Pilot Study
Brief Title: GLP-1s to Enhance Lasting Optimal Weight
Acronym: GLOW
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00127025
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Obesity
Keywords: Weight Loss; Muscle Loss; Physical Disability; Bone Density; Older Adults
MeSH Terms: conditions — Obesity; Weight Loss; Muscular Atrophy | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tirzepatide (Experimental): Tirzepatide injection once weekly for 9 months
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Tirzepatide will be initiated at a dose of 2.5 mg weekly and increased as tolerated to 5 mg weekly at four weeks for the remainder of the 9-month intervention period. Participants who are unable to tolerate the 5 mg dose will be decreased to the 2.5 mg dose.
  Other Names: Zepbound

SUMMARY:
The goal of this study is to examine how tirzepatide affects body composition, bone health, and physical performance in older adults over a nine-month period. Participants will take tirzepatide weekly, have clinic visits every 4 weeks, meet study doctor and registered dietitian every 4 weeks in person or video conference, attend group intervention sessions twice a month via video conference, weigh daily with a study-provided smart scale, keep a record of all foods and beverages consumed, and use a study-provided activity tracker to keep track of daily step counts.

DETAILED DESCRIPTION:
This study will enroll 40 older adults with obesity (or overweight with a weight-related comorbidity) in a 9-month pilot to examine the effects of tirzepatide on body composition, bone health, and physical performance. All participants will receive tirzepatide, 5 mg per week and counseling sessions (group and individual) on diet quality and physical activity as well as behavioral strategies to facilitate dietary and physical activity changes. Participants will be expected to weigh themselves daily on a smart scale, record their food and beverage consumption, and keep track of daily step counts over the 9-month intervention period. Body composition, bone health, and physical performance will be measured at baseline prior to intervention and approximately nine months later. This data will be used to examine the effects of tirzepatide on total and appendicular lean and total fat mass measured by DXA; hip and spine bone mineral density measured by DXA; and leg strength and physical performance (expanded Short Physical Performance Battery, 400-m walk).

ELIGIBILITY:
Inclusion Criteria:

* BMI 30-37 kg/m2 or BMI 27-<30 kg/m2 with at least 1 weight-related comorbidity
* community dwelling
* able to provide own transportation to study visits
* willing to provide informed consent
* willing to take terzepatide for 9 months
* agree to all study procedures/assessments
* approved for participation by the study physician

Exclusion Criteria:

* dependent on a cane or walker or needing assistance with any activity of daily living
* history of mild cognitive impairment or dementia or cognitive impairment on Montreal Cognitive Assessment (MoCA score <22)
* evidence of depressive symptoms (Center for Epidemiologic Studies Depression scale score =>16
* use of >1 tobacco product/day or 4/week or vaped >1/week in past year
* excessive alcohol use in past month (>7 drinks/week for women; >14 drinks/week for men)
* weight loss or gain >5% in past 3 months
* vegan or other severe dietary restriction
* history of binge eating disorder
* regular participation in high intensity aerobic or resistance exercise training >150 mins/week
* severe arthritis, fracture, chronic injury, or other musculoskeletal disorder that prevents walking independently
* joint replacement or other orthopedic surgery in past 6 months or planned in next 12 months
* osteoporosis (self report or DXA t-score <= -2.5 on total hip and/or femoral neck)
* uncontrolled hypertension (systolic >160 OR diastolic >100 mmHg) upon repeated assessments
* type 1 diabetes
* uncontrolled type 2 diabetes (HbA1c >7.5%), type 2 diabetes diagnosed within last year, or newly identified type 2 diabetes (HbA1c >6.5%)
* dialysis or abnormal kidney function (eGFR <30 ml/min/1.73m2)
* liver disease or abnormal liver function (ALT levels 2 times above normal limit)
* severe anemia (Hb <11 g/dL)
* potassium or sodium above or below normal limits
* uncontrolled thyroid disease (hypo/hyper) or requiring recent (past 3 months) adjustments in thyroid hormone supplementation or TSH <0.45 or >4.5 mU/L
* stroke, heart attack, heart failure hospitalization, or revascularization procedure within the past year; New York heart failure Class >2; COPD requiring oxygen use; uncontrolled angina; PAD diagnosis within the last year; progressive neurologic disease (e.g., Parkinson's, ALS, MS); other diseases suggesting a life-expectancy <3 years
* personal or family history of medullary thyroid carcinoma, history of multiple endocrine neoplasia syndrome type 2, or any other cancer (except non-melanoma skin cancers) requiring treatment in past year
* history of gastroparesis or pancreatitis
* cholelithiasis, severe irritable bowel syndrome or Crohn's disease
* history of stomach or small intestinal surgery (except appendectomy but including surgery for weight loss)
* recent (within 4 weeks) acute respiratory illness including influenza, COVID-19
* overnight hospitalization within the past 6 months
* regular use of growth hormones, medications prescribed for weight management, prescription osteoporosis medications, certain prescription medications for diabetes including insulin, sulfonylurea, meglitinides, GLP-1 agonists, SGLT2 inhibitors
* use of oral steroids for >1 month within the last 3 months
* current participation in another intervention research study
* planned out of town trips greater than 3 weeks in the next year

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in total body lean mass | Baseline to Month 9
  Change in total body lean mass will be measured by DXA scan
Change in appendicular lean mass | Baseline to Month 9
  Change in appendicular lean mass will be measured by DXA scan
Change in total body fat mass | Baseline to Month 9
  Change in total body fat mass will be measured by DXA scan
Change in total hip bone mineral density | Baseline to Month 9
  Change in total hip bone mineral density will be measured by DXA scan
Change in lumbar spine bone mineral density | Baseline to Month 9
  Change in lumbar spine bone mineral density will be measured by DXA scan
Change in 400 meter walk time | Baseline to Month 9
  Change in the time it takes to walk 400 meters (10 laps on an indoor, 20-meter course). The 400 meter walk is a test of exercise tolerance and aerobic fitness.
Change in lower extremity physical performance score | Baseline to Month 9
  Change in lower extremity physical performance will be assessed by the expanded Short Physical Performance Battery. Activities include side-by-side, semi-tandem, tandem and one leg stand balance tests; 4 meter walk; 4 meter narrow walk; and time to rise from a chair five times. Total score ranges from 0-4 with higher scores indicating better lower extremity physical performance.
Change in leg strength | Baseline to Month 9
  Change in leg extensor strength will be assessed using the Keiser AIR300 Leg Press System.

SECONDARY OUTCOMES:
Change in thigh intramuscular fat tissue | Baseline to Month 9
  Change in thigh intramuscular fat tissue will be measured by CT scan
Change in thigh muscle volume | Baseline to Month 9
  Change in thigh muscle volume will be measured by CT scan
Change in total skeletal muscle mass | Baseline to Month 9
  Change in total skeletal muscle mass will be assessed by D3 creatine
Change in total volumetric bone mineral density of the hip | Baseline to Month 9
  Change in total volumetric bone mineral density of the hip will be measured by CT scan
Change in hip bone strength | Baseline to Month 9
  Change in hip bone strength will be measured by CT scan
Change in total volumetric bone mineral density of the radius | Baseline to Month 9
  Change in total volumetric bone mineral density of the radius will be measured by high-resolution peripheral quantitative CT
Change in total volumetric bone mineral density of the tibia | Baseline to Month 9
  Change in total volumetric bone mineral density of the tibia will be measured by high-resolution peripheral quantitative CT
Change in c-telopeptide of type 1 collagen (CTX) | Baseline to Month 9
  Change in c-telopeptide of type 1 collagen (CTX) will be measured by enzyme-linked immunosorbent assay
Change in procollagen type 1 n-terminal propeptide (P1NP) | Baseline to Month 9
  Change in procollagen type 1 n-terminal propeptide (P1NP) will be measured by enzyme-linked immunosorbent assay
Change in bone-specific alkaline phosphatase (BALP) | Baseline to Month 9
  Change in bone-specific alkaline phosphatase (BALP) will be measured by enzyme-linked immunosorbent assay
Change in osteocalcin | Baseline to Month 9
  Change in osteocalcin will be measured by enzyme-linked immunosorbent assay

CONTACTS AND LOCATIONS:
Overall Officials: Denise Houston, PhD, Principal Investigator — Atrium Health Wake Forest Baptist
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No